CLINICAL TRIAL: NCT02868684
Title: Multi-modality Magnetic Resonance Imaging Biomarkers of Mild Traumatic Brain Injury: a Longitudinal Cohort Study
Brief Title: Imaging Biomarkers of Mild Traumatic Brain Injury: a Longitudinal Cohort Study
Status: Completed | Type: Observational
Sponsor: First Affiliated Hospital Xi'an Jiaotong University (Other)
Collaborators: Second Affiliated Hospital of Wenzhou Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: NSFC81571752-1
Record Dates: First submitted 2016-08-09; First posted 2016-08-16 (Estimated); Last update posted 2022-05-12 (Actual); Status verified 2022-05

CONDITIONS: Mild Traumatic Brain Injury; Posttraumatic Stress Disorder; Affective and Somatic Complaints; Cognitive Impairments
MeSH Terms: conditions — Brain Concussion; Stress Disorders, Post-Traumatic; Cognitive Dysfunction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- mild traumatic brain injury
- Healthy controls

SUMMARY:
This longitudinal cohort study aims to detect the topographical nature of the white matter microstructure and resting state functional connectivity patterns across the whole brain in the evolution of pathology as a function of time following mild TBI. All consecutively patients with the non-contrast head CT because of acute head trauma from the local emergency department (ED) formed the initial population of this study. Age, sex, education-level matched healthy controls will also be enrolled. The initial scan will performed within 7 days post-injury. Clinical assessment was performed within 24 hours of MR imaging and included a broad neuropsychological and symptom assessments. Follow-up examination will conduct at 1 month, 3 month, 6-12 months.

ELIGIBILITY:
Inclusion Criteria:

* Glasgow Coma Score of 13-15;
* one or more of the following: loss of consciousness (if present) < 30 min, post-traumatic amnesia (if present) < 24 h, and/or other transient neurological abnormalities such as focal signs, seizure, and intracranial lesion not requiring surgery.
* no contraindications to MRI;
* injury within 7 days;
* agreement to communicate by telephone or e-mail for 1, 3 to 6-12 months after enrollment and come back to the hospital for follow-up

Exclusion Criteria:

* history of neurological disease
* head injury, or history of substance or alcohol abuse, intubation and/or presence of a skull fracture
* administration of sedatives on arrival in the emergency department
* spinal cord injury, manifestation of mild TBI due to other injuries (e.g., systemic injuries, facial injuries, or intubation) or other problems (e.g., psychological trauma, language barrier, or coexisting medical conditions), or caused by penetrating craniocerebral injury.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All consecutively patients with the non-contrast head CT because of acute head trauma from the local emergency department (ED) formed the initial population of this study. Three research assistants (trained, board-certified neurologist or neurosurgeon) monitored the ED and hospital wards on a daily basis to identify new admissions. Screening for mild traumatic brain injury (TBI) was based on the World Health Organization's Collaborating Centre for Neurotrauma Task Force.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2016-08 (Actual); Primary Completion 2020-08 (Actual); Study Completion 2020-09 (Actual)

PRIMARY OUTCOMES:
Correlation between brain diffusion tensor imaging measures and Posttraumatic Stress Disorder symptom | 1 month

SECONDARY OUTCOMES:
Changes in post-concussive symptoms | baseline, 1 month
changes in affective complaints | baseline and follow-up
Changes in somatic complaints | baseline and follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Ming Zhang, M.D, Principal Investigator — First Affiliated Hospital Xi'an Jiaotong University
Locations (1):
- First Affiliated Hospital of Xi'an Jiaotong University, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Niu X, Bai L, Sun Y, Wang Y, Bai G, Yin B, Wang S, Gan S, Jia X, Liu H. Mild traumatic brain injury is associated with effect of inflammation on structural changes of default mode network in those developing chronic pain. J Headache Pain. 2020 Nov 23;21(1):135. doi: 10.1186/s10194-020-01201-7. PMID 33228537